CLINICAL TRIAL: NCT03354793
Title: Impact of Endometriosis on the Risk of Obstetric Complications in Spontaneous Pregnancy: a Multicentric Italian Study
Brief Title: Endometriosis and Risk of Obstetric Complications
Status: Completed | Type: Observational
Sponsor: Endometriosis Treatment Italian Club (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor
Other Study IDs: ETIC002
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Endometriosis; Pregnancy Complications
MeSH Terms: conditions — Endometriosis; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometriosis: Survey on first pregnancy after endometriosis diagnosis
  Interventions: Other: Survey on first pregnancy after endometriosis diagnosis
- non endometriosis: Survey on first pregnancy
  Interventions: Other: Survey on first pregnancy

INTERVENTIONS:
Other: Survey on first pregnancy after endometriosis diagnosis — Obstetric complications were noted
  Groups: endometriosis
Other: Survey on first pregnancy — Obstetric complications were noted
  Groups: non endometriosis

SUMMARY:
The aim of this study is to compare the rate of obstetric complications at first spontaneous pregnancy among women with endometriosis, with the rate of obstetric complications at first spontaneous pregnancy among women without endometriosis

DETAILED DESCRIPTION:
All women followed up for a surgical or clinical/sonographic diagnosis of endometriosis in 11 italian referral Centres for the treatment of endometriosis, completed a questionnaire regarding their previous pregnancies. The same questionnaire was completed by women, attending a routine gynecologic visit, in whom surgery or clinical/sonographic evaluation excluded endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 50 years old women with at least one previous spontaneous pregnancy > 12 weeks with surgical or clinical/sonographic diagnosis of endometriosis or in whom surgical or clinical/sonographic evaluation ruled out endometriosis

Exclusion Criteria:

* Pregnancy achieved by assisted reproductive techniques
* Pregnancy terminated before 12 gestational weeks
* Twin pregnancy
* Preexisting hypertension
* Lupus like anti-coagulant
* Non corrected uterine malformation
* Recurrent abortion

Ages: 30 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: All continuous women attending endometriosis clinics or undergoing a routine gynecological examination matching the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 844 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Pre-term delivery | 2 years
  comparison of rate of preterm delivery in the two groups

SECONDARY OUTCOMES:
Placenta praevia | 2 years
  comparison of rate of placenta praevia in the two groups

OTHER OUTCOMES:
Intra uterine Growth Restriction | 2 years
  comparison of rate of IUGR fetuses in the two groups
HELLP syndrome | 2 years
  comparison of rate of HELLP syndrome in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Berlanda, MD, Principal Investigator — Endometriosis Treatment Italian Club

REFERENCES:
- [Derived] Berlanda N, Alio W, Angioni S, Bergamini V, Bonin C, Boracchi P, Candiani M, Centini G, D'Alterio MN, Del Forno S, Donati A, Dridi D, Incandela D, Lazzeri L, Maiorana A, Mattei A, Ottolina J, Orenti A, Perandini A, Perelli F, Piacenti I, Pino I, Porpora MG, Scaramuzzino S, Seracchioli R, Solima E, Somigliana E, Venturella R, Vercellini P, Vigano P, Vignali M, Zullo F, Zupi E; Endometriosis Treatment Italian Club (ETIC). Impact of endometriosis on obstetric outcome after natural conception: a multicenter Italian study. Arch Gynecol Obstet. 2022 Jan;305(1):149-157. doi: 10.1007/s00404-021-06243-z. Epub 2021 Oct 8. PMID 34623489